CLINICAL TRIAL: NCT02591719
Title: Effects of Repetitive Transcranial Magnetic Stimulation Based on Neural Activation in Language Performance in Stroke Patients With Non-fluent Aphasia
Brief Title: Effects of rTMS Based on Neural Activation in Language Performance in Stroke Patients With Non-fluent Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1507-308-006/P2
Record Dates: First submitted 2015-10-22; First posted 2015-10-29 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Aphasia
Keywords: Functional Near-Infrared Spectroscopy; Stroke; Aphasia; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MagPro magnetic stimulator (HF rTMS) (Experimental): Most activated area from fNIRS with language task: Perilesional Broca's area
  Interventions: Device: MagPro magnetic stimulator (HF rTMS)
- MagPro magnetic stimulator (sham) (Sham Comparator): Most activated area from fNIRS with language task: Perilesional Broca's area
  Interventions: Device: MagPro magnetic stimulator (sham)
- MagPro magnetic stimulator (LF rTMS) (Active Comparator): Most activated area from fNIRS with language task: Contralesional homologs of Broca's area
  Interventions: Device: MagPro magnetic stimulator (LF rTMS)

INTERVENTIONS:
Device: MagPro magnetic stimulator (HF rTMS) — Most activated area from fNIRS findings: Perilesional Broca's area. Use the true coil. High frequency rTMS (10Hz), Number of total stimuli: 800, Location: perilesional Broca's area, Intensity: 100% of resting motor threshold, Coil orientation: tangential to scalp, in combination with speech therapy(35-40min) after each rTMS session, Daily 10 treatment session
  Other Names: High frequency rTMS
  Arms: MagPro magnetic stimulator (HF rTMS)
Device: MagPro magnetic stimulator (sham) — Most activated area from fNIRS findings: Perilesional Broca's area. Use the sham coil. High frequency rTMS (10Hz), Number of total stimuli: 800, Location: perilesional Broca's area, Intensity: 100% of resting motor threshold, Coil orientation: tangential to scalp, in combination with speech therapy(35-40min) after each rTMS session, Daily 10 treatment session
  Other Names: Sham stimulation
  Arms: MagPro magnetic stimulator (sham)
Device: MagPro magnetic stimulator (LF rTMS) — Most activated area from fNIRS findings: Contralesional homologs of Broca's area.
  Use the true coil. Low frequency rTMS (1Hz), Number of total stimuli: 1200, Location: Contralesional homologs of Broca's area (Pars triangularis), Intensity: 90% of resting motor threshold, Coil orientation: tangential to scalp, in combination with speech therapy(35-40min) after each rTMS session, Daily 10 treatment session
  Other Names: low frequency rTMS
  Arms: MagPro magnetic stimulator (LF rTMS)

SUMMARY:
The aim of this study is to assess the safety and clinical efficacy of repetitive transcranial magnetic stimulation (rTMS) based on hemodynamic brain activity pattern with functional near infrared spectroscopy (fNIRS) in early poststroke nonfluent aphasia patients.

DETAILED DESCRIPTION:
Most conventional rTMS studies employed an inhibitory low frequency protocol for the contralesional homologs of Broca's area.

In the present randomized controlled trial, investigators will perform fNIRS prior to rTMS treatment to select the stimulation method. Stimulation site (perilesional or contralesional) and frequency (excitatory high or inhibitory low) will be determined by activation pattern from the fNIRS with language task in individual patients.

The patient who shows a dominant neural activity at perilesional Broca's area on fNIRS scanning will be randomly allocated into two groups: high frequency stimulation group and sham stimulation group. If a patient shows a dominant neural activity at contralesional homologs of Broca's area on fNIRS scanning, the patient will be allocated to a low frequency stimulation group.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 yrs old
* Right-handed
* Radiologically confirmed left hemisphere stroke within 6 months
* Fluent in Korean
* First ever stroke
* Non-fluent (motor-dominant) aphasia
* Written informed consent

Exclusion Criteria:

* Previous medical histories of stroke, cerebral vascular operation,
* Seizure
* Patients with traumatic brain injury
* Unable to perform the language task
* Severe cognitive impairment (MMSE less than 16)
* Skin lesion in the stimulation site of scalp
* Metal implants in the body (cardiac pacemaker or aneurysm clip)
* Pregnancy, breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
BNT (Boston Naming Test) | up to 2 weeks
  speech evaluation tool for measuring the confrontational word retrieval function

SECONDARY OUTCOMES:
WAB (Western Aphasia Battery;speech evaluation tool for screening the presence, degree, and type of aphasia) | up to 6 weeks
  Baseline(when allocated to each study arm), after the completion of 10 session of 'rTMS+speech therapy' (that is, 2 weeks later from the baseline), 4 weeks later after the completion of 10 session of 'rTMS+speech therapy'
LI (Laterality Index; From fNIRS findings, LI=L-R/L+R (L and R represent maximum or mean left and Right hemispheric HbO (oxyhemoglobin) or total Hb values, respectively) | up to 6 weeks
  Baseline(when allocated to each study arm), after the completion of 10 session of 'rTMS+speech therapy' (that is, 2 weeks later from the baseline), 4 weeks later after the completion of 10 session of 'rTMS+speech therapy'
BNT (Boston Naming Test) | 4 weeks
  speech evaluation tool for measuring the confrontational word retrieval function

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam-si, Korea, Gyeonggi-do, South Korea